CLINICAL TRIAL: NCT07090707
Title: Prospective Exploratory Phase II Study of PD-1 Inhibitor Therapy Versus Radiotherapy in MPR Patients After Neoadjuvant Immunochemotherapy for Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: PD-1 Inhibitor Therapy Versus Radiotherapy in MPR Patients With Locally Advanced HNSCC After Neoadjuvant Immunochemotherapy (HNC-SYSU-006)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-1094-02
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: HNSCC; PD-1; Radiotherapy
Keywords: HNSCC; PD-1; radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1（PD-1） (Experimental): Radiotherapy free treatment: the experimental group took PD-1 inhibitor maintenance regimen.
  Interventions: Drug: PD-1inhibitor
- Arm 2（radiotherapy） (Active Comparator): conventional radiotherapy (chemoradiotherapy) regimen, and received comprehensive treatment according to the guidelines (radiotherapy or platinum-based concurrent chemoradiotherapy as stipulated in the guidelines).
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: PD-1inhibitor — The PD-1 monoclonal antibody was the same as the neoadjuvant therapy before surgery, and the postoperative level was maintained at Q3*6.
  Arms: Arm 1（PD-1）
Radiation: radiotherapy — According to the guidelines, concurrent chemoradiotherapy is required, and carboplatin (50mg/m2) plus concurrent radiotherapy or cisplatin (30mg/m2) plus concurrent radiotherapy is optional.
  Arms: Arm 2（radiotherapy）

SUMMARY:
Head and neck malignant tumors rank as the sixth most common type of malignancy worldwide, with approximately 90% being squamous cell carcinoma (Head and Neck Squamous Cell Carcinoma, HNSCC). Globally, there are about 650,000 new cases of HNSCC annually, with China contributing approximately 350,000 new cases each year. At initial diagnosis, 60% of patients already present with locally advanced HNSCC, necessitating comprehensive treatment strategies.

In the first half of the 20th century, radiotherapy was the primary treatment for HNSCC. However, due to its relatively low local control rate (70%), high rate of distant metastasis (20%), and low 5-year overall survival (OS) rate (40%), coupled with significant early and late adverse effects, radiotherapy often brought severe challenges to patients. For instance, 95% of patients developed radiation-induced oral mucositis, nearly all experienced xerostomia, taste disorders, radiation-induced dental caries, restricted mouth opening, swallowing difficulties, aspiration, and other functional impairments. Some patients even suffered severe complications, with 6% developing radiation-induced osteonecrosis of the jaw, and 0.1% experiencing secondary cancers such as radiation-induced sarcoma or squamous cell carcinoma in the head and neck region. Other complications, such as radiation-induced encephalopathy, also posed significant threats to patients' safety and quality of life. As surgical techniques improved towards the end of the 20th century, surgery gradually replaced radiotherapy as the dominant treatment for HNSCC.

Over the past four decades, despite the use of comprehensive treatments based on surgery supplemented by radiotherapy, chemotherapy, and targeted therapy, the 5-year survival rate for locally advanced HNSCC has not significantly improved, remaining around 50%. Recently, with the advent of immunotherapy centered on PD-1 inhibitors, treatment outcomes for HNSCC patients have improved markedly, and the therapeutic landscape is undergoing significant transformation. Concurrently, many studies have focused on neoadjuvant immunotherapy prior to surgery. In locally advanced lung cancer, neoadjuvant chemoimmunotherapy has been proven safe and effective through phase III clinical trials. Similarly, studies on head and neck tumors have shown that neoadjuvant immunotherapy-whether PD-1 monotherapy or in combination with chemotherapy-demonstrates favorable safety and efficacy. However, for patients who respond well to immunochemotherapy and achieve pathological downstaging, how to evaluate the relationship between therapeutic efficacy, staging, and prognosis, as well as how to plan subsequent treatments, remains unclear in existing guidelines. For some patients with locally advanced HNSCC who achieve major pathological response (MPR) or pathological complete response (pCR) after neoadjuvant immunochemotherapy and undergo extensive primary tumor resection and thorough neck lymph node dissection, there is no research to clarify whether postoperative adjuvant radiotherapy based on pretreatment TNM staging is still necessary.

Some studies suggest that for patients with pN1 stage, adjuvant radiotherapy after thorough neck lymph node dissection does not significantly impact local control or long-term survival. Literature indicates that the recurrence rate of cervical lymph nodes in N1-stage head and neck squamous cell carcinoma is approximately 8%, meaning that about 92% of N1-stage patients who receive postoperative radiotherapy to the cervical lymphatic drainage area might be overtreated. For patients who achieve pCR after neoadjuvant immunochemotherapy, continuing radiotherapy in the original region after high-quality surgery further increases the likelihood of overtreatment. For locally advanced HNSCC patients who achieve pCR or MPR in the primary tumor and lymph nodes, whether routine radiotherapy should be administered following high-quality surgical resection and lymph node dissection remains controversial in the academic community.

This leads to our clinical question: In patients with locally advanced HNSCC who achieve MPR in both the primary tumor and lymph nodes after neoadjuvant immunochemotherapy and undergo standard surgical treatment, can maintenance therapy with PD-1 inhibitors replace adjuvant radiotherapy?

This study aims to enroll patients who have undergone neoadjuvant immunochemotherapy followed by standard surgical treatment and achieved MPR in both the primary tumor and lymph nodes. Patients will be divided into an experimental group and a control group. The experimental group will receive maintenance therapy with PD-1 inhibitors, while the control group will follow guideline-recommended adjuvant treatments (radiotherapy or concurrent chemoradiotherapy based on platinum compounds) according to tumor classification and staging before neoadjuvant immunochemotherapy. Outcomes such as 2-year

ELIGIBILITY:
Inclusion Criteria:

* In this study, patients with locally advanced head and neck squamous cell carcinoma (AJCC 8th) who underwent standard surgical treatment after neoadjuvant immunochemotherapy and showed MPR in both primary lesions and lymph node pathology were selected. Locally advanced squamous cell carcinoma of head and neck includes: i) T3, N0, M0; 2) T1-T3, N1-N2, M0; 3) T4a, N0-2, M0.
* No history of other malignant tumors
* Ages 18-75
* Normal baseline inspection:

  1. The absolute value of neutrophil granulocyte (ANC) ≥1.5x109/L in the last 14 days without the use of granulocyte colony stimulating factor;
  2. Platelets ≥100×109/L without blood transfusion in the past 14 days;
  3. Hemoglobin &gt without blood transfusion or use of erythropoietin within the last 14 days; 9g/dL;
  4. Total bilirubin ≤1.5× upper limit of normal value (ULN);
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN in patients with liver metastasis);
  6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
  7. Good coagulation function, defined as International Standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. Subjects whose baseline TSH is outside the normal range can be enrolled if total T3 (or FT3) and FT4 are within the normal range;
  9. The myocardial enzyme profile was within the normal range (if the researchers comprehensively judged that the simple laboratory abnormality was not clinically significant, it was also allowed to be included);
  10. For female subjects of childbearing age, a urine or serum pregnancy test should be tested negative within 3 days prior to receiving the first study drug administration (day 1 of Cycle 1). If the urine pregnancy test results cannot be confirmed negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy;
  11. If there is a risk of conception, all subjects (male or female) shall use contraception with an annual failure rate of less than 1% for the entire duration of treatment up to 120 days after the last study drug administration (or 180 days after the last chemotherapeutic drug administration).

  5 Sign informed consent

Exclusion Criteria:

* 1 HNSCC is not the initial diagnosis of other malignant tumors or neoadjuvant therapy.
* Prior to treatment An active autoimmune immune disease requiring systemic therapy (e.g. the use of disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred in the last 2 years. Alternative therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1) HBV viral load &lt before initial administration; At 1000 copies /ml (200 IU/ml), subjects should receive anti-HBV therapy to avoid viral reactivation throughout the study treatment period 2) For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required

* Active HCV infected subjects (HCV antibody positive and HCV-RNA level above the lower limit);
* Pregnant or lactating women;
* The presence of any serious or uncontrolled systemic disease, such as:

  1. The resting electrocardiogram (ECG) presents significant and severely uncontrollable abnormalities in rhythm, conduction or morphology, such as complete left bundle branch block, Ⅱ degree or above heart block, ventricular arrhythmia or atrial fibrillation;
  2. Unstable angina pectoris, congestive heart failure, and NYHA grade ≥ 2 chronic heart failure;
  3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before treatment;
  4. Poor blood pressure control (systolic > 140 mmHg, diastolic > 90 mmHg);
  5. A history of non-infectious pneumonia requiring glucocorticoid therapy or clinically active interstitial lung disease within 1 year prior to initial administration;
  6. Active pulmonary tuberculosis;
  7. There is an active or uncontrolled infection that requires systemic treatment;
  8. Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
  11. Urine routine indicated urine protein ≥++, and confirmed 24 hours urine protein quantity > 1.0 g;
  12. Patients with mental disorders and unable to cooperate with treatment;
* Medical history or evidence of disease that may interfere with test results, prevent subjects from fully participating in the study, abnormal values of treatment or laboratory tests, or other conditions that the investigator considers unsuitable for enrollment. The investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival （DFS） | 2 years
  DFS(by months) is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease DFS is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease relapse.
Percentage of adverse events graded by CTCAE v5.0 and RTOG | 90 days after surgery
  Percentage of adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0) and RTOG. Change From Baseline 90 days after surgery.

SECONDARY OUTCOMES:
Overall survival(OS) | 5 years
  The time(measured by months) from day 1 of study treatment until death from any cause.
regional recurrence-free survival (RRFS) | 2 years
  The time( by months) from randomization to clinically confirmed recurrence in the lymph node drainage area. Deaths were counted in RRFS.
distant metastasis free survival (DMFS) | 2 years
  The time( by months) from randomization to clinically confirmed distant metastasis.
Number and percentage of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 and RTOG | 2 years
  The detail number and percentage of adverse events by every systems Assessed by CTCAE v5.0 and RTOG.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No